

| BI Study Number: | 0135-0348 |
|---|---|
| Title: | Characteristics and in-hospital outcomes of Chinese elderly (>80 years) patients with acute ischemic stroke receiving intravenous recombinant tissue plasminogen activator treatment within 4.5 hours of symptom onset |
| NCT number: | NCT05395351 |
| Date: | January 28, 2022 |

This page has been added to the Statistical and Epidemiological Analysis Plan (SEAP) to reflect the requirements by ClinicalTrials.gov. This information is not part of the standard document.



## STATISTICAL AND EPIDEMIOLOGICAL ANALYSIS PLAN (SEAP) FOR NON-INTERVENTIONAL STUDIES (NIS)

| Document Number: | c37691036-01 |
|---|---|
| BI Study Number: | 0135-0348 |
| BI Investigational<br>Product(s) | Actilyse® (Alteplase) |
| Title: | Characteristics and in-hospital outcomes of Chinese elderly (>80 years) patients with acute ischemic stroke receiving intravenous recombinant tissue plasminogen activator treatment within 4.5 hours of symptom onset |
| Brief lay title: | Alteplase in elderly AIS during hospitalization |
| SEAP version identifier: | 1.0 |
| Date of last version of SEAP: | |
| NIS Statistician | |
| [SEAP author] | |
| NIS | |
| [SEAP reviewer] | |
| NIS Data | |
| [SEAP reviewer] | |

**Proprietary confidential information** 

© 2021 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

| I. IADLE CUNTENTS | 1. | <b>TABLE</b> | CONTENTS |
|-------------------|----|--------------|----------|
|-------------------|----|--------------|----------|

| TITI | LE PAG | E |
|------|--------|---------------------------------------------------|
| 1. | TABL | E CONTENTS |
| 2. | LIST | OF ABBREVIATIONS |
| 3. | RESPO | ONSIBLE PARTIES |
| 4. | PURPO | OSE AND SCOPE |
| 5. | AMEN | IDMENTS AND UPDATES |
| 6. | RESEA | ARCH QUESTION AND OBJECTIVE |
| 7. | RESEA | ARCH METHODS |
| 7.1 | STU | JDY DESIGN9 |
| 7.2 | SET | TING |
| 7.3 | STU | JDY POPULATION |
| 7.4 | STU | JDY VISITS |
| 8. | VARIA | ABLES |
| 8.1 | EXI | POSURES 12 |
| 8.2 | OU' | TCOMES |
| 8 | 3.2.1 | Primary outcomes |
| 8 | 3.2.2 | Secondary outcomes |
| 8.3 | | VARIATES |
| 9. | | SOURCES |
| 10. | | MANAGEMENT AND SOFTWARE/TOOLS |
| 10. | | FTWARE/TOOLS |
| 10.2 | | NDLING OF MISSING VALUES |
| | | NDLING OF INCONSISTENCIES IN DATA AND OUTLIERS 15 |
| 11. | | ANALYSIS |
| 11. | 1 MA | IN ANALYSIS |
| | 1.1.1 | Primary outcomes |
| 1 | 1.1.2 | Second outcomes |
| 11.3 | 3 SAI | FETY ANALYSIS |
| 12. | QUAL | ITY CONTROL 19 |

| Statistical and Epidemiological Analysis Plan (SEAP) for Non- | c37691036-01 |
|---|---|
| Interventional Studies (NIS) Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affili | |
| Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affil | liated companies |
| 13.1 PUBLISHED REFERENCES | 20 |
| 13.2 UNPUBLISHED REFERENCES | 20 |
| ANNEX 1. ADDITIONAL INFORMATION | 21 |
| 1. DEFINITION OF VARIABLES | 21 |
| 2. DICTIONARY OF VARIABLES | 22 |
| 3. MOCK TABLE&FIGURE | 22 |
| ANNEY 2 DEVIEWEDS AND ADDROVAL SIGNATURES | 36 |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

AIS Acute Ischemic Stroke

ASD Absolute Standardized Difference

BI Boehringer Ingelheim CI Confidence Intervals

CSA Chinese Stroke Association CSCA Chinese Stroke Centre Alliance

EVT Endovascular Treatment IQR Interquartile Range

IV Intravenous

IVT Intravenous Thrombolysis

NIHSS National Institutes of Health Stroke Scale

NIS Non-interventional Study

NIS-DMRP Non-interventional Study-data Management and Review Plan

RCTs Randomized Controlled Trials

rt-PA Recombinant Tissue Plasminogen Activator

RWE Real-world Evidence

SEAP Statistical and Epidemiological Analysis Plan

SOPs Standard Operation Procedures
TIA Transient Ischemic Attack

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. RESPONSIBLE PARTIES

NIS Statistician [SEAP author]

| SEAP | reviewers are: |
|---------|----------------|
| | BI NIS |
| • | NIS Data |
| • | RWE |
| • | TSTAT |
| NA<br>• | TM Epi |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. PURPOSE AND SCOPE

Using the Chinese Stroke Centre Alliance (CSCA) data to describe the in-hospital clinical outcomes regarding safety and effectiveness for AIS patients who were treated with IV rt-PA within 4.5 hours of symptom onset, aged above 80 years, as well as between 18 and 80 years. We plan to apply and incorporate the results of this study (providing in-hospital outcomes), together with another non-interventional study in China (providing 1-year clinical outcomes), as well as results from randomized controlled trials conducted in other countries, to support local label update: to remove the age restriction (>80 years) from the label of Actilyse in China.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. AMENDMENTS AND UPDATES

Not applicable.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. RESEARCH QUESTION AND OBJECTIVE

**Research question:** What are the in-hospital clinical outcomes among Chinese AIS patients, who were treated with IV rt-PA within 4.5 hours of symptom onset in different age groups (18 to 80 years and above 80 years).

#### **Primary objective:**

• To describe the all-cause mortality during hospitalization of AIS patients who were treated with IV rt-PA within 4.5 hours of symptom onset, among those aged 18 to 80 years and >80 years, respectively.

#### **Secondary objectives:**

- To describe other in-hospital clinical outcomes (including proportion of patients with hemorrhagic stroke during hospitalization, change of NIHSS score from before IV rt-PA treatment to 24 hours after IV rt-PA treatment, mRS score at discharge, proportion of patients with stroke recurrence during hospitalization, and length of hospitalization) of AIS patients who were treated with IV rt-PA within 4.5 hours of symptom onset, among those aged 18 to 80 years and >80 years, respectively.
- To describe the characteristics of AIS patients who arrived or were admitted to the hospital within 4.5 hours of symptom onset and were treated with or without IV rt-PA among different age groups (18 to 80 years and above 80 years).
- To describe the percentage of patients receiving IV rt-PA treatment within 4.5 hours of symptom onset among AIS patients aged 18 to 80 years and above 80 years who arrived at or were admitted to the hospital within 4.5 hours of symptom onset.



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RESEARCH METHODS

#### 7.1 STUDY DESIGN

This is a non-interventional study based on existing data from CSCA platform.

### **Patient groups:**

Patients in this study will be divided into 4 groups:

- Group 1: AIS patients aged >80 years who received IV rt-PA within 4.5 hours of symptom onset
- Group 2: AIS patients aged 18 to 80 years who received IV rt-PA within 4.5 hours of symptom onset
- Group 3: AIS patients aged >80 years who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive thrombolysis treatment
- Group 4: AIS patients aged 18 to 80 years who arrived or were admitted to the hospital within 4.5 hours of symptom onset and did not receive thrombolysis treatment

The baseline characteristics will be described in groups 1 to 4.

The clinical outcomes during hospitalization will be observed in groups 1 to 2.

In addition, the percentage of AIS patients who received IV rt-PA treatment within 4.5 hours of onset will be calculated among 4.5 hours hospital arrival AIS patients, and IVT eligible patients (3.5 hours hospital arrival or admission and without IVT absolute contraindication), in each age group of 18 to 80 years and >80 years, respectively.

In China, rt-PA is only indicated in AIS patients aged 18 to 80 years. Therefore, it is possible that AIS patients aged >80 years who received IV rt-PA are different from other patients in terms of their baseline characteristics (channeling). To evaluate the potential channeling, in this study we will compare the baseline characteristics of AIS patients aged >80 years treated with IV rt-PA within 4.5 hours of symptom onset (Group 1) with those in Group 2 and Group 3.



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The flow of data selection for each of the 4 reporting patient groups is depicted in <u>Figure 1</u> below.

Primary outcome

All-cause mortality during hospitalization of patients in groups 1 and 2. Secondary outcomes Proportion of patients with hemorrhagic stroke during hospitalizatio
 Change of NIHSS score from before IV rt-PA treatment to 24 hours after IV rt-PA treatment mRS score at discharge.

Proportion of patients with stroke recurrence during hospitaliza Inclusion Criteria Length of hospitalization; Aged >80 years Group 1 All the above in-hospital secondary outcomes will be observed in Group I from Aug. 2015 to Jul. 2019 Percentage of iv rt-PA treatment among AIS patients arrived or were Aged 18-80 year ≥18 years old Group 2 admitted to the hospital within 4.5 hours of symptom onset; Diagnosed as AIS at admission Percentage of iv n-PA treatment within 4.5 hours of symptom onset among eligible AIS patients (3.5-hour arrival or admission);
 The percentage of IV n-PA treatment will be calculated based on age Patients with Arrived at or be admitted into hospital within 4.5 hours of groups (18-80 years and > 80 year). Baseline characteristics of each group;
 Differences in baseline characteristics of patients in group 1 compared symptom onset For patients in the is rt-PA groups only: received iv rt-PA within 4.5 hours of with group 2 and group 3. Aged >80 years Group 3 symptom onset Did not receive thrombolysis treatment Aged 18-80 year Group 4 Exclusion Criteria · With documented IVT absolute contraindication except age to IV rt-PA treatment according to the SmPC. Key data missing (age, gender, baseline NIHSS, time of symptom onset, IVT treated or not, time of iv alteplase treatment)

• Received thrombolysis agents other than iv rt-PA (urokinase, teneeteplase, recombinant plasminogen activator, prourokinase, streptokinase) Received endovascular treatment
 Received iv rt-PA after 4.5 hours of symptom onset

Figure 1 Patient groups for the non-interventional study

Note: AIS, Acute Ischemic Stroke; CSCA, Chinese Stroke Centre Alliance; iv, Intravenous; rt-PA, Recombinant Tissue Plasminogen Activator; IVT, Intravenous Thrombolysis.

#### 7.2 SETTING

In this study, AIS patients from 1476 hospitals (720 Grade 2 hospitals and 756 Grade 3 hospitals) in the CSCA platform from Aug 2015 to Jul 2019 will be used.

#### 7.3 STUDY POPULATION

Acute ischemic stroke (AIS) patients who were treated with IV rt-PA or did not receive thrombolysis treatment within 4.5 hours of symptom onset, aged ≥18 years old.

No sampling will be undertaken and all patients who meet all the inclusion criteria and none of the exclusion criteria will be included.

The inclusion and exclusion criteria are listed below:

#### Inclusion Criteria:

- Patient registered in the CSCA platform from Aug 2015 to Jul 2019
- ≥18 years old
- Diagnosed as AIS at admission
- Arrived or admitted into hospital within 4.5 hours of symptom onset

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• For patients in the iv rt-PA groups only: received IV rt-PA within 4.5 hours of symptom onset.

#### **Exclusion Criteria:**

- Documented IVT absolute contraindication
- Key data missing (age, gender, baseline National Institutes of Health Stroke Scale [NIHSS], time of symptom onset, IVT treated or not, time of IV alteplase treatment)
- Received thrombolysis agents other than IV rt-PA (urokinase, tenecteplase, recombinant plasminogen activator, prourokinase, streptokinase)
- Received endovascular treatment
- Received IV rt-PA after 4.5 hours of symptom onset.

#### 7.4 STUDY VISITS

Not applicable.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. VARIABLES

#### 8.1 EXPOSURES

The exposure in this study is the use of IV rt-PA among AIS patients within 4.5 hours of symptom onset.

#### 8.2 OUTCOMES

### 8.2.1 Primary outcomes

All-cause mortality during hospitalization of patients in Group 1 and Group 2.

#### 8.2.2 Secondary outcomes

- Proportion of patients with hemorrhagic stroke during hospitalization
- Change of NIHSS score from before IV rt-PA treatment to 24 hours after IV rt-PA treatment
- mRS score at discharge
- Proportion of patients with stroke recurrence during hospitalization
- Length of hospitalization

All the above in-hospital secondary outcomes will be observed in Group 1 and Group 2.

- Percentage of IV rt-PA treatment among AIS patients arrived or were admitted to the hospital within 4.5 hours of symptom onset
- Percentage of IV rt-PA treatment within 4.5 hours of symptom onset among eligible AIS patients (3.5-hour arrival or admission)

The percentage of IV rt-PA treatment will be calculated based on age groups (18-80 years and > 80 year).



#### 8.3 COVARIATES

Covariates include the following variables at baseline:

- Age
- Gender (male, female)
- Stroke severity (baseline NIHSS)
- Time from symptom onset to hospital arrival or admission
- Smoking (current smoker, former smoker, never smoker)

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Alcohol consumption (yes, no)
- Comorbidities at baseline (diabetes, prior coronary heart disease /myocardial infarction, atrial fibrillation/flutter, prior heart failure, carotid stenosis, peripheral vascular disease, prior stroke/transient ischemic attack(TIA), hypertension, dyslipidaemia)
- Comedication at baseline (antiplatelet, anticoagulation, antidiabetics, antihypertensive drug, lipid-lowering drug)
- For IV rt-PA treated patients:
  - a) Time from symptom onset to treatment
  - b) Time from hospital arrival or admission to treatment (door-to-needle time)
  - c) Dosage of rt-PA
- For No IV rt-PA treated patients:
  - a) Reasons for not being treated with IV rt-PA
- Education (primary school or below, junior high school, senior high school, junior college or above)
- Medical insurance status (urban employee basic medical insurance, urban resident basic medical insurance, new rural cooperative medical insurance, other medical insurance, no insurance)
- Hospital level (Grade 2, Grade 3).

Variables collected during hospitalization:

- Lab values: blood-glucose, C-reactive protein;
- Clinical symptoms: evaluation of swallowing ability, pneumonia;

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. DATA SOURCES

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. DATA MANAGEMENT AND SOFTWARE/TOOLS

Routine operations of the CSCA are conducted and managed by the CSA staff. These operations are as follows: update and maintain the CSCA web-based data collection and management tool; develop and run site feedback reports and execute research analyses as part of its role as the CSCA data coordinating centre. The CSCA's data coordinating centre resides at the

#### 10.1 SOFTWARE/TOOLS

All statistical analyses were performed using SAS Version 9.4 software. All ASD>10 were considered significant.

#### 10.2 HANDLING OF MISSING VALUES

Every reasonable attempt have been undertaken to ensure completeness of data collection. In general, missing data will be treated as missing. No data imputation will be performed for the missing data. Due to the nature of existing data, the interpretation is based on non-missing data.

#### 10.3 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS

Missing and erroneous values in patient cases can significantly impact the ability to perform research for identifying risk factors and disease distribution, treatment progression. This study is mainly based on review of data collected from CSCA and aims at evaluating differences in clinical practice of IV-rtPA treatment among AIS patients from 2015 to 2019. Data follow-up period has already been finished. Thus, data cannot meet the criteria of this study will be excluded.

#### Exclusion criteria:

- 1. Missing key data including
- Contraindications to venous thrombolysis within a time window
- symptom onset time (or last known well time);
- baseline NIHSS;
- whether received IVT treatment or not;
- the time of IVT treatment (For patients in the IV rt-PA groups only);
- Received thrombolysis agents other than IV rt-PA (Urokinase);
- Received endovascular treatment:
- Received IV rt-PA after 4.5 hours of symptom onset (For patients in the IV rt-PA groups only):
- age and gender
- 2. Contradiction of time period:
  - IVT treatment time earlier than symptom onset time (or last known well time);
  - treatment time earlier than hospital arrival time;
  - hospital arrival time earlier than symptom onset time

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

3. Diagnosed with intracranial hemorrhage (ICH), Transient Ischemic Attack (TIA), subarachnoid hemorrhage (SAH), or unspecific stroke

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11. DATA ANALYSIS

The study is descriptive in nature. The calculation will be based on the available data. Selected outcomes will be analyzed with data from hospital participated in CSCA. Selected outcomes will also be standardized by hospital (based on CSCA).

For continuous data, descriptive statistics (number of patients, mean, standard deviation [SD], minimum, median, interquartile range, and maximum) will be presented. Categorical data will be presented as frequency and proportion with 95% CI as appropriate.

#### 11.1 MAIN ANALYSIS

The baseline characteristics (covariates) as listed in Section 8.3 will be analysed by using descriptive statistics for all 4 groups in this study, where Group 1 is compared against group 2 and Group 1 is compared against Group 3 to evaluate the potential channeling. Absolute standardized difference (ASD) between the compared groups will be calculated, in which a ≥10% ASD will be considered a meaningful difference.

The primary outcome is the all-cause mortality during hospitalization. The primary outcome will be described using descriptive statistics for Group 1 and Group 2. The secondary outcome as listed in Section 8.2.2 will also be described using descriptive statistics for Group 1 and Group 2. Additionally, if the baseline characteristics of patients in group 1 are comparable to patients in group 3 (ASD<10%), then we will describe the in-hospital outcomes for group 3 patients, including all-cause mortality during hospitalization, proportion of patients with hemorrhagic stroke during hospitalization, mRS score at discharge, proportion of patients with stroke recurrence during hospitalization, and length of hospitalization. If the baseline characteristics of patients in group 1 and group 3 are not comparable, then we will not describe the above outcomes in group 3.

For general statistical considerations, the descriptive statistics for continuous variables will include mean, standard deviation, or median, interquartile range (IQR); for categorical variables, counts, percentages, and 95% CI will be included. For categorical variables, 95% Clopper-Pearson confidence interval will be used.

In terms of the display of decimal places, mean, median, and IQR will be reported to one more decimal place than the raw data recorded in the database. Standard deviation and 95% confidence interval will be reported to two more decimal places than the raw data recorded in the database. P-value will be reported to fourth decimal place if available.

### 11.1.1 Primary outcomes

All-cause mortality during hospitalization of patients in Group 1 and Group 2 (Table 1)

• Proportion of died AIS patients during hospitalization who were treated with IV rt-PA within 4.5 hours of symptom onset among those aged 18 to 80 years(Group 2) and >80 years(Group 1);

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.1.2 Second outcomes

# Among all AIS patients during hospitalization who were treated with IV rt-PA within 4.5 hours of symptom onset (patients Group 1 and Group 2) (Table 2)

- Proportion of patients with hemorrhagic stroke during hospitalization
- Change of NIHSS score from before IV rt-PA treatment to 24 hours after IV rt-PA treatment
- mRS score at discharge
  - a) Discharge MRS score classification
  - b) Discharge MRS score (0-1)
- Proportion of patients with stroke recurrence during hospitalization
- Length of hospitalization;

# Among all AIS patients during hospitalization on 18-80 years age groups (Group 2 and Group 4) and > 80 year age groups (Group 1 and Group 3)(Table 3)

- Percentage of IV rt-PA treatment among AIS patients arrived or were admitted to the hospital within 4.5 hours of symptom onset
- Percentage of IV rt-PA treatment within 4.5 hours of symptom onset among eligible AIS patients (3.5-hour arrival or admission)



#### 11.3 SAFETY ANALYSIS

This is a NIS based on existing data. From safety information collecting and reporting perspective, this study will not involve individual medical record review, thus no adverse event/adverse drug reaction information is required to collect.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 12. QUALITY CONTROL

The quality control, review, and monitoring plan are summarized below. Greater details are documented in the NIS-DMRP.

The study will strictly follow BI standard operation procedures (SOPs). In addition, this study will follow key elements of the Guideline for GPP The statistical analytic approach will be reviewed/repeated by a second analyst. The study report will be reviewed, approved and archived per BI SOP.

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

13. REFERENCES

13.1 PUBLISHED REFERENCES

NA

13.2 UNPUBLISHED REFERENCES

NA

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ANNEX 1. ADDITIONAL INFORMATION**

**Type** 

#### 1. DEFINITION OF VARIABLES

- (1) Patients characteristics
  - --Smoke including current smoking & cessation of smoking within previous year
- (2) Medical history

Variable Name

- --DM including self-reported history of diabetes or current use of hypoglycemic drugs
- --Hypertension including self-reported history of hypertension or current use of antihypertensive drugs

Label & Value

| | 1 | mid | -14 | n ! |
|---|---|---|---|---|
| | | pid | character | Patient ID |
| | 2 | hunitID | character | Hospital ID |
| | 3 | Hlevel | numerical | Hospital Grade |
| | 4 | hname | character | Hospital Name |
| | 5 | gender | numerical | Gender:1=Male;2=Female |
| | 6 | Agen | numerical | Age At Admission |
| | 7 | d_diag | character | Final diagnosis: |
| | | | | 1= Ischemic stroke;2=TIA;3=ICH;4=SAH;5=Other |
| | | A_NIHSSn | numerical | Fisrt Time Nihss After Hospital Arrival |
| | 9 | H_SMK | numerical | History Of Smoke: 1-never smoker; 2- former smoker; 3- |
| | | | | current smoker; other-unclear): |
| | 10 | H_DRINK | numerical | History Of Drink (Including Past Habit of Drinking But Not In Last Year; Or Still Drinking) :0=No;1=Yes |
| | 11 | H_DM1 | numerical | History Of Diabetes: Selfreport History or Medication Use: |
| | 12 | Н НҮРТ1 | m11m ami a a 1 | 0=No;1=Yes<br>History Of Hypertentsion: Selfreport History or Medication Use: |
| | 12 | п_птгт | numerical | 0=No;1=Yes |
| | 13 | Stt lipid | numerical | History Of Hypelipidemia: Selfreport History or Medication Use: |
| | | _ • | | 0=No;1=Yes |
| | 14 | H_AFIB | character | History of atrial Fibrillation: 0=No;1=Yes |
| | 15 | H_HF | character | History of heart failure: 0=No;1=Yes |
| | 16 | H_CHDMI | numerical | History of chronic heart disease or Myocardial Infarction: 0=No;1=Yes |
| | 17 | H_PVD | character | History of peripheral vascular disease: 0=No;1=Yes |
| | 18 | H_CSTENO | character | History of carotid artery stenosis: 0=No;1=Yes |
| | 19 | H StrokeTIA | numerical | History of stroke or TIA |
| | 20 | onset_door_time | numerical | Hours from onset to hospital arrival |
| | 21 | onset_needle_time | numerical | Hours from onset to rt-PA Treatment |
| | 22 | Door needle time | numerical | Hours from hospital arrival to rt-PA Treatment |
| | 23 | TPA | numerical | Treatment with Tpa: 0=No;1=Yes |
| | 24 | H_PLT | character | History of medication of Antiplatelet agent: 0=No;1=Yes |
| | 25 | H COAG | character | History of medication of Anticoagulant drugs: 0=No;1=Yes |
| | 26 | TPA_R | character | Reasons for not being treated with IV rt-PA:1= Beyond the rt-PA |
| | | | | intravenous thrombolysis time window;2= ontraindications to |
| | | | | intravenous thrombolysis within a time window;3= Hospital |
| | | | | related or other reasons;4= Economic reasons;5= The patient or family refused; other=unclear. |
| | 27 | DYS RESULTFMT | numerical | 1= Function good;0 or 2= Function of difficult; other=unclear |
| Ι. | - ' | | | 1 1 unction good, o of 2—1 unction of difficult, other—uncidal |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

| Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | |
|---|---|---|
| Variable Name | Type | Label & Value |
| 28 EDUcat | numerical | 1=college;2=high school;3=below elementary; other=unclear |
| 29 Insurance | | 1=UEBMI;4=URBMI;5=NRCMS;6=Self-pay; other=other |
| | | medical insurance |
| 30 I_FGn | numerical | blood-glucose |
| 31 I_CRP_UNITn | numerical | C-reactive protein |
| | Variable Name 28 EDUcat 29 Insurance 30 I_FGn | Variable Name 28 EDUcat 29 Insurance Type numerical character 30 I_FGn numerical |

- --CHD or MI including Chronic Heart Disease or self-report history of myocardial infarction
- --AF including self-report history of Atrial fibrillation
- --Previous stroke including self-report history of ischemic stroke, intracranial hemorrhage or subarachnoid hemorrhage
- --TIA including self-report history of transient ischemic attack
- --Dyslipidaemia including self-report history of lipid metabolism disorders or current use of lipid-lowering drugs

#### 2. DICTIONARY OF VARIABLES

#### 3. MOCK TABLE&FIGURE

Primary outcomes:

Table 1. All-cause mortality during hospitalization of patients in Group 1 and Group 2.

| Variables | Group 1 (N= [%]) | Group 2 (N= [%]) |
|---------------------|------------------|------------------|
| All-cause mortality | n (%) (95%CI) | n (%) (95%CI) |

Secondary outcomes:

Table 2. Secondary outcomes during hospitalization of patients in Group 1 and Group 2.

| Variables | Group 1 (N= [%]) | Group 2 (N= [%]) |
|---|---|---|
| Proportion of patients with hemorrhagic stroke | | |
| during hospitalization | n (%) (95%CI) | n (%) (95%CI) |
| Change of NIHSS score from before IV rt-PA | | |
| treatment to 24 hours after IV rt-PA treatments | | |
| | Nmiss (%) | Nmiss (%) |
| | Mean±SD | Mean±SD |
| | Min-Max | Min-Max |
| | Median (IQR) | Median (IQR) |
| mRS score at discharge | | |
| Discharge mRS score classification | | |
| Missing | n (%) (95%CI) | n (%) (95%CI) |
| 0 | n (%) (95%CI) | n (%) (95%CI) |
| 1 | n (%) (95%CI) | n (%) (95%CI) |
| 2 | n (%) (95%CI) | n (%) (95%CI) |
| 3 | n (%) (95%CI) | n (%) (95%CI) |
| 4 | n (%) (95%CI) | n (%) (95%CI) |
| 5 | n (%) (95%CI) | n (%) (95%CI) |
| Discharge mRS score (0-1) | n (%) (95%CI) | n (%) (95%CI) |

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

| prietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | |
|---|---|---|
| Variables | Group 1 (N= [%]) | Group 2 (N= [%]) |
| Proportion of patients with stroke recurrence | e | |
| during hospitalization | n (%) (95%CI) | n (%) (95%CI) |
| Length of hospitalization, d | Nmiss (%) | Nmiss (%) |
| • | Mean±SD | $Mean\pm SD$ |
| | Min-Max | Min-Max |
| | Median (IQR) | Median (IQR) |

Table 3. Proportion of 4.5 h IV-rtPA treatment among all AIS patients (arrived or admitted within 4.5 hours of symptom onset) based on age groups & Proportion of 4.5h IV-rtPA treatment among 3.5h IVT eligible patients.

| | | > 80 years (N= |
|----------------------------------|----------------------|----------------|
| Proportion | 18-80 years (N= [%]) | [%]) |
| 4.5h IV-rtPA / all AIS patients | n (%) (95%CI) | n (%) (95%CI) |
| 4.5h IV-rtPA / 3.5h IVT eligible | n (%) (95%CI) | n (%) (95%CI) |



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

| Treprietary termital | entiter information o 2021 Boen | iringer ingemenn internation | ar dinerr or one or more or it | s arrinated companies |
|---|---|---|---|---|

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

| Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

| - | Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 



Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)

c37691036-01 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS) c37691036-01 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 2. REVIEWERS AND APPROVAL SIGNATURES

The NIS SEAP must be sent for review to the following individuals **prior to approval**.

| Reviewer | NIS involving BI<br>product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi* | X | X | X |
| NIS Data Manager | X | X | X |
| TSTAT<br>(for NISnd only) | X | X | X |
| RWE CoE | X | X | |

<sup>\*</sup> When BI NIS lead is not TM Epi

**Study Title:** Characteristics and in-hospital outcomes of Chinese elderly (>80 years) patients with acute ischemic stroke receiving intravenous recombinant tissue plasminogen activator treatment within 4.5 hours of symptom onset

**Study Number: 0135-0348** 

Name/Date:

Protocol Version:1.0

Position:

I herewith certify that I agree to the content of the study SEAP and to all documents referenced in the study SEAP.

| Position: | Name/Date: | Signature: |
|-----------|------------|------------|
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |

Signature: